CLINICAL TRIAL: NCT04718857
Title: The Construction and Empirical Research of Hospital Chronic Disease Health Management Information Platform From the Perspective of Internet
Brief Title: Chronic Disease Health Management Information Platform
Status: Withdrawn | Type: Observational
Why Stopped: Intervention change
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-701
Record Dates: First submitted 2020-12-03; First posted 2021-01-22 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Online education — health education

SUMMARY:
Based on the combination of domestic and foreign experience and the needs of patients as the orientation, this research gives full play to the hospital's advantages in chronic disease management, and uses network information technology to develop a systematic and intelligent system that integrates prevention, diagnosis and treatment, follow-up, and education.

DETAILED DESCRIPTION:
Patients with hypertension are showing a trend of getting younger and younger, and high-normal blood pressure is increasing rapidly among the young and middle-aged people aged less than 65 years.

Young and middle-aged patients with hypertension have a lower absolute short-term cardiovascular risk, but their lifetime risk is higher.

Studies have shown that the awareness rate, treatment rate and control rate ("three rates") of young and middle-aged hypertensive patients in my country need to be improved urgently.

Improving the knowledge and behavior of young and middle-aged hypertensive patients with disease, treatment compliance and self-health management has become the focus of research.

"Internet + medical" through information network technology, innovative service models have become a trend.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 to 59 years old according to the World Health Organization (WHO) age classification criteria, meet the diagnostic criteria for hypertension published in the "Guidelines for the Prevention and Control of Hypertension in China", and are diagnosed with essential hypertension;
* Patients are conscious and possess Normal reading, comprehension and expression skills;
* use a smart phone to surf the Internet and send and receive information, accept and use the outpatient chronic disease health management platform services;
* Informed consent, voluntarily participate in this research.

Exclusion Criteria:

* Patients with severe organic heart disease and other cardiovascular and cerebrovascular diseases;
* Chronic liver and kidney failure;
* Patients with malignant tumors;
* Persons who have participated in other forms of Internet + health management.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Young and middle-aged patients with essential hypertension in the Cardiovascular Outpatient Department of a tertiary A general hospital
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Health literacy level | 1 YEAR
  The individual's ability to acquire, understand, evaluate and exchange information in different environments throughout the life process to improve, maintain and improve health
Self-management behavior ability | 1 YEAR
  The self-management behavior assessment scale for hypertensive patients includes six dimensions of medication management, condition monitoring, diet management, exercise management, rest and work management, and emotional management, as well as the assessment of the total level of self-management. There are 33 items in total, the sum of the scores of each item For the final total score of the scale, the items use Likert 5-level scoring method, which is always (5 points), often (4 points), sometimes (3 points), rarely (2 points), never (1 point).
Blood pressure compliance rate | 1 YEAR
  The "Guidelines for the Prevention and Treatment of Hypertension in China (2018 Revised Edition)" recommends that blood pressure be reduced to <140/90 mmHg. In this study, the blood pressure compliance rate means that the patient's blood pressure measurement value is less than 140/90mmHg and stable for more than one month. Blood pressure compliance rate = number of people meeting blood pressure/total number of people receiving chronic disease management in outpatient clinics * 100%.

CONTACTS AND LOCATIONS:
Overall Officials: FANG LIANGYU, Study Director — Outpatient Department of the Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Outpatient Department of the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No